CLINICAL TRIAL: NCT03327272
Title: Impact of Local Steroid Application in Extreme Lateral Lumbar Interbody Fusion
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not enroll, PI decided not to proceed.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kern Singh, Professor, Department of Orthopaedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17102301
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stenosis; Herniated Nucleus Pulposus; Degenerative Disc Disease; Spondylosis; Myelopathy; Radiculopathy; Myeloradiculopathy
MeSH Terms: conditions — Constriction, Pathologic; Intervertebral Disc Degeneration; Spondylosis; Spinal Cord Diseases; Radiculopathy | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Local injection of methylprednisolone (Active Comparator): Drug: methylprednisolone Injection of 80mg methylprednisolone injectable suspension at surgical site prior to incision closure
  Interventions: Drug: Methylprednisolone
- Local injection of saline (Placebo Comparator): Administration of saline at surgical site prior to incision closure.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Methylprednisolone — Injection of 80mg Depomedrol injectable suspension at surgical site prior to incision closure
  Other Names: Depomedrol
  Arms: Local injection of methylprednisolone
Drug: Saline — Administration of saline at surgical site prior to incision closure
  Arms: Local injection of saline

SUMMARY:
Neural injury is a well-known complication following extreme lateral lumbar interbody fusion (XLIF). It has been found that up to 9.4% of patients will have either temporary or persistent neurologic deficit. This occurs with traversal of the psoas muscle or direct injury to lumbosacral plexus or sympathetic ganglion. While often temporary, it can cause hip flexor weakness, thigh numbness, or pain.

Several studies have demonstrated reduced patient reported pain scores following steroid administration, particularly in the early postoperative period. However, few studies have investigated the efficacy of intraoperative local injection of corticosteroid in reducing the incidence and duration of postoperative pain or neurologic injury for XLIF patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the incidence and duration of postoperative pain is reduced in the subjects receiving a local injection of methylprednisolone when compared to placebo following XLIF.

The investigators hypothesize that subjects undergoing XLIF who receive local methylprednisolone will have:

1. Reduced incidence and duration of postoperative pain and neurologic injury
2. Shorter hospital stay
3. Better short- and long-term outcomes

The study also aims to answer the following questions:

1. Do subjects who receive local corticosteroids have a reduced incidence and duration of postoperative pain and neurologic deficit compared to those who receive placebo?
2. Do subjects who receive local corticosteroids have a reduced hospital stay compared to those who received placebo?
3. Is local corticosteroid therapy associated with improved short and long-term outcomes?

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a 1- to 2-level XLIF
* Diagnosis: myelopathy, radiculopathy, myeloradiculopathy, stenosis, herniated nucleus pulposus, degenerative disc disease, spondylosis, osteophytic complexes, and foraminal stenosis
* Patients able to provide informed consent

Exclusion Criteria:

* Allergies or other contraindications to medicines in the protocol including:
* Existing history of gastrointestinal bleeding
* Lumbar spine trauma
* Unable to speak, read, or understand English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 2 year postoperative
  Change in Visual Analogue Scale (VAS) Back and Leg pain score from preoperative value will be assessed. VAS back and leg pain scores assess pain in each region on a scale from 0-10 with 0 being no pain and 10 being worst pain imaginable.

SECONDARY OUTCOMES:
Physical Functioning | 2 year postoperative
  Patient-Reported Outcomes Measurement Information System (PROMIS) physical function score as compared to preoperative value. This score assesses physical function and is scaled from 0-100 with 100 indicating greater functioning and 0 indicating worse functioning.
Disability | 2 year postoperative
  Oswestry Disability Index (ODI) score as compared to preoperative score. ODI assesses disability out of a total of 50 points and is scaled to a percentage of total possible points with 0 indicating no disability and 100 indicating severe disability.
General health status | 2 year postoperative
  Short Form (SF)-12 Survey scores as compared to preoperative values. SF-12 assesses general physical and mental health on a scale of 0 to 100 with higher scores indicating superior health status
Narcotic Consumption | 2 year postoperative
  The total amount of narcotic use for each subject will be recorded. Dosages of narcotics will be converted to morphine equivalents
Length of Stay | 1 week postoperative
  The number of hours of hospitalization from entering the recovery room (time zero) until patient meets discharge criteria
Post-operative adverse events | 1 week postoperative
  Post-operative nausea and vomiting, Gastro-esophageal reflux, Ileus, Venous thromboembolic events, Respiratory depression/airway compromise, Renal insufficiency, Wound Complications, Admission to the ICU

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No